CLINICAL TRIAL: NCT00006263
Title: Phase II Trial of Temozolomide, Carboplatin and Neupogen in High-Grade Gliomas, Both Newly-Diagnosed and Recurrent
Brief Title: Carboplatin, Temozolomide, and Filgrastim in Treating Patients With Newly Diagnosed or Recurrent High-Grade Glioma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068203; NYU-0004H; NYU-0029H; NCI-G00-1856
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult brain stem glioma; adult glioblastoma; childhood high-grade cerebral astrocytoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma | interventions — Filgrastim; Carboplatin; Temozolomide

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combining carboplatin, temozolomide, and filgrastim in treating patients who have newly diagnosed or recurrent high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with newly diagnosed high-grade glioma treated with temozolomide, carboplatin, and filgrastim (G-CSF).
* Determine the toxicity of this treatment regimen in these patients.
* Determine the rate of tumor progression in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to disease category (glioblastoma multiforme vs anaplastic astrocytoma vs several other high-grade mixed gliomas).

Patients receive carboplatin IV over 4 hours on days 1-2; oral temozolomide every 12 hours on days 1-5; and filgrastim (G-CSF) subcutaneously or IV daily starting no earlier than day 7 and continuing until blood counts recover. Treatment repeats every 28 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 102-222 (17-37 per each of 6 strata) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed glioblastoma multiforme or anaplastic astrocytoma

  * Residual tumor on postoperative MRI
* Bidimensionally measurable disease

PATIENT CHARACTERISTICS:

Age:

* Under 65

Performance status:

* Karnofsky or Lansky 70-100% OR
* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Hemoglobin at least 8 g/dL (transfusion allowed)
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGPT no greater than 3 times ULN

Renal:

* Age 5 years and under: Creatinine less than 1.2 mg/dL
* Age over 5 to 10 years: Creatinine less than 1.5 mg/dL
* Age over 10 to 15 years: Creatinine less than 1.8 mg/dL
* Age over 15 years: Creatinine less than 2.4 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months

Other:

* No other concurrent serious medical condition that would preclude study
* Able to tolerate oral medications
* No prior malignancy for which patient received prior chemotherapy or spinal irradiation
* No history of severe allergic reaction to platinum-containing compounds
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 72 hours since prior filgrastim (G-CSF)

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent steroids for tumor-related cerebral edema allowed
* No concurrent corticosteroids for solely antiemetic purposes

Radiotherapy:

* No prior or concurrent radiotherapy

Surgery:

* Recovered from prior surgery
* No concurrent surgery

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 1997-11

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L. Finlay, MB, ChB, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States